CLINICAL TRIAL: NCT05887726
Title: A Single-arm, Prospective Clinical Study on the Antitumor Activity and Safety of Zanubrutinib Combined With R-CHOP Regimen in the Treatment of Newly Diagnosed DLBCL With High-risk Factors
Brief Title: Zanubrutinib Combined With R-CHOP Regimen in the Treatment of Newly Diagnosed DLBCL With High-risk Factors
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Liaoning Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZR-CHOP HR
Record Dates: First submitted 2023-03-20; First posted 2023-06-05 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-02

CONDITIONS: Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — zanubrutinib; Rituximab; Cyclophosphamide; Epirubicin; Vincristine; Prednisone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Zanubrutinib + R-CHOP (Experimental)
  Interventions: Drug: Zanubrutinib; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Epirubicin; Drug: Vincristine; Drug: Prednisone

INTERVENTIONS:
Drug: Zanubrutinib — Zanubrutinib 160mg bid p.o d0-d20(21-day cycles)
Drug: Rituximab — Rituximab 375 mg/m2 i.v d0(21-day cycles)
Drug: Cyclophosphamide — Cyclophosphamide 750 mg/m2 i.v d1(21-day cycles)
Drug: Epirubicin — Epirubicin 75 mg/m2 i.v d1 or liposome adriamycin 35mg/m2 i.v d1(21-day cycles)
Drug: Vincristine — Vincristine 1.4 mg/m2 i.v d1 (2 mg max) (21-day cycles)
Drug: Prednisone — Prednisone 100 mg p.o d1-d5 (21-day cycles)

SUMMARY:
This study is a prospective, open-label, single-arm phase II clinical study to evaluate the safety and efficacy of zanubrutinib plus R-CHOP (ZR-CHOP) as the first-line therapy for newly diagnosed diffuse large B-cell lymphoma patients with high-risk factors.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed DLBCL patients have one of the following risk factors(including but not limited to double expression, extranodal involvement, high ki67, bulky)；
2. Age ≥ 18 years old;
3. At least one measurable lesion (defined as lymph node lesion ≥15mm, extra-segmental lesions ≥ 10mm);
4. ECOG performance status 0-2;
5. Functions of major organs meet the following conditions: Echocardiography left ventricular ejection fraction ≥50%; Creatinine clearance ≥30 ml/min; ALT and AST≤3 times the normal range；
6. Hematopoietic function should meet the following conditions: Platelet count ≥50×109/L; Hemoglobin ≥ 8.0g /dL; Absolute count of neutrophil (ANC)≥1.0×109/L;
7. Expected survival of ≧3 months

Exclusion Criteria:

1. Major surgery within 4 weeks before treatment;
2. Severe organ dysfunction(including but not limited to complications of uncontrolled cardiovascular diseases, blood clotting disorders, connective tissue diseases, serious infectious diseases and other diseases);
3. Patients who cannot cooperate with treatment or follow-up on time.
4. Pregnant or lactating females;
5. any uncontrolled active systemic infection requiring intravenous (IV) antibiotics;
6. There was a history of other active malignant diseases within the 2 years prior to study entry, except for: (1) adequately treated cervical carcinoma in situ; (2) local skin basal cell carcinoma or squamous cell carcinoma; (3) previous malignant disease that is under control and has undergone local radical treatment (surgical or other forms).
7. History of severe hemorrhagic disorders, such as hemophilia A, hemophilia B, von Willebrand's disease, or spontaneous bleeding requiring blood transfusion or other medical intervention
8. Human immunodeficiency virus (HIV) infection or the following serological status reflecting the presence of active hepatitis B or C virus infection: a. Hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) are present. Patients who are HBCAB-positive, HBsAg negative, have no hepatitis b virus (HBV) DNA (< 20 IU/mL), and agree to be monitored for HBV virus reactivation can be enrolled. Antibodies to the hepatitis C virus (HCV) are present. HCV antibody-positive patients with no HCV RNA detected could be included in the group.
9. The presence of any life-threatening disease, medical condition, or organ system dysfunction that the investigator believes may affect the subject's safety or pose a risk to the study.
10. The researchers think it is not suitable to participate in this experiment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Complete response rate（CRR） | Up to approximately 2.5 years

SECONDARY OUTCOMES:
Overall response rate （ORR） | Up to approximately 2.5 years
Progression-free Survival(PFS) | Up to approximately 2.5 years
Overall survival (OS) | Up to approximately 2.5 years
Duration of Response | At 2 years
Incidence of adverse event | At 2 years
Assessment of the correlation between MYD88、CD79B、NOTCH1、BCL6、NOTCH2 or other gene abnormality and efficacy. | At 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojing Xing, Ph.D, Principal Investigator — Liaoning Cancer Hospital & Institute
Locations (1):
- Xing Xiaojing, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No